CLINICAL TRIAL: NCT06257628
Title: MACE CDS Software Master Enrollment Protocol
Status: Withdrawn | Type: Observational
Why Stopped: Business decision
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2.7.2.1
Record Dates: First submitted 2023-10-18; First posted 2024-02-14 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Events
Keywords: Emergency Department; Major Adverse Cardiac Events
MeSH Terms: conditions — Cardiovascular Diseases; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Index Event: Patients with at least one Beckman High Sensitivity Troponin test at the Emergency Department visit
  Interventions: Device: Index Event

INTERVENTIONS:
Device: Index Event — Patients with at least one Beckman High Sensitivity Troponin test at the Emergency Department visit

SUMMARY:
This protocol will collect real world EHR data to support the product development life cycle activities associated with developing the Major Adverse Cardiac Events (MACE) Clinical Decision Support (CDS) software.

The data will also be utilized in subsequent clinical validation to support an FDA application and/or applications to other regulatory agencies as needed.

DETAILED DESCRIPTION:
The primary objective is to develop a machine learning tool which predicts risk of 30-day MACE (major adverse cardiac event) risk stratification among patients visiting ED with suspicion of ACS (Acute Coronary Syndrome).

The data will also be utilized in subsequent clinical validation. In addition to retrospective Electronic Health Record (EHR) data, Health Information Exchange (HIE) data and patient reported outcomes will be collected to capture 30-day MACE outcomes, as applicable.

ELIGIBILITY:
Inclusion Criteria:

* All genders, races, ethnicities

Exclusion Criteria:

* ≤ 18 years old presenting to the ED and for clinical validation only, adults < 22 years old

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients visiting ED with suspicion of Acute Coronary Syndrome (ACS).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Performance Characteristics NPV (Negative Predictive Value), Specificity and Sensitivity | Within 30-days from the Emergency Department Visit with suspicion of ACS (Acute Coronary Syndrome)
  Clinical performance of MACE (Major Adverse Cardiac Events) CDS (Clinical Decision Support) tool to identify a patient's risk of for having a MACE (Major Adverse Cardiac Events) within 30 days, with both a single High-Sensitive Troponin and a second High-Sensitive Troponin (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Drain, Study Director — Beckman Coulter
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Kettering Health, Kettering, Ohio